CLINICAL TRIAL: NCT05880225
Title: Musical Rhythm Sensitivity to Scaffold Social Engagement in Autism Spectrum Disorder
Brief Title: Reciprocal Imitation Training and Musical Rhythm Sensitivity in Autistic Toddlers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Miriam Lense, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH123029
Record Dates: First submitted 2023-05-10; First posted 2023-05-30 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; imitation; social communication; rhythm; music
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reciprocal Imitation Training (RIT) (Active Comparator): Children (n=20) receive 30 sessions of Reciprocal Imitation Training (RIT), delivered in 40-60 minute sessions 2-3 times/week.
  Interventions: Behavioral: Reciprocal Imitation Training
- Music-Enhanced Reciprocal Imitation Training (meRIT) (Experimental): Children (n=20) receive 30 sessions of music-enhanced Reciprocal Imitation Training (meRIT), delivered in 40-60 minute sessions 2-3 times/week.
  Interventions: Behavioral: music-enhanced Reciprocal Imitation Training

INTERVENTIONS:
Behavioral: Reciprocal Imitation Training — As a naturalistic developmental behavioral intervention (NDBI), Reciprocal Imitation Training (RIT) utilizes contingent imitation, linguistic mapping, modeling, prompting, and contingent reinforcement to train object and gesture imitation during play activities.
  Arms: Reciprocal Imitation Training (RIT)
Behavioral: music-enhanced Reciprocal Imitation Training — Music-enhanced imitation training uses music and rhythm to enhance the predictability and salience of the strategies utilized within the Reciprocal Imitation Training platform (i.e., contingent imitation, linguistic mapping, modeling, prompting, and contingent reinforcement to train object and gesture imitation during play activities).
  Arms: Music-Enhanced Reciprocal Imitation Training (meRIT)

SUMMARY:
The primary goal of this study is to examine rhythm sensitivity as a predictor of response to naturalistic developmental behavioral intervention (NDBIs) in autistic toddlers. Toddlers receive either Reciprocal Imitation Training (RIT), an evidence-based NDBI that supports children's imitation and social communication skills, or a music-enhanced version of RIT. Throughout their participation in the intervention, toddlers will complete study procedures of viewing naturalistic videos of infant-directed singing and other social scenes while eye gaze data is collected.

DETAILED DESCRIPTION:
Social communication makes use of predictable, rhythmic behaviors and children are sensitive to the rhythm of social interaction from infancy. The goal of the current study is to investigate if social rhythm sensitivity, measured via children' entrained eye-looking when viewing videos of infant-directed singing, predicts autistic toddlers' response to naturalistic developmental behavioral intervention (NDBI). Following eligibility testing and baseline assessments, children are randomized to receive either 30 sessions of Reciprocal Imitation Training (RIT), an NDBI that uses evidence-based strategies to support children's imitation and social communication development, or a music-enhanced version of RIT that embeds music and rhythm within the RIT platform (meRIT). Children's imitation skills are assessed before and after the intervention programs. Children's rhythm sensitivity is assessed via repeated eye-tracking sessions throughout baseline, intervention, and two-weeks after the intervention ends.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of autism / autism spectrum disorder
* 18-36 months of age

Exclusion Criteria:

* Major hearing or visual impairment (e.g., congenital nystagmus), seizure disorder, genetic syndromes, or gestational age <=34 weeks.

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in rhythmically entrained eye-looking (eye-tracking) | Change from baseline through 2-week follow-up post-intervention
  Trajectories of rhythmically entrained eye-looking to predictable and unpredictable child-directed singing assessed via passive eye-tracking.

SECONDARY OUTCOMES:
Change in overall fixation to eyes (eye-tracking) | Change from baseline through 2-week follow-up post-intervention
  Trajectories of proportion of time spent fixating on the eyes while viewing predictable and unpredictable child-directed singing assessed via passive eye-tracking.
Change in child elicited motor imitation | Change from baseline to 2-weeks follow-up after intervention
  Children's performance on the Motor Imitation Scale (score 0-32). Higher scores indicate greater performance.
Change in child spontaneous motor imitation | Change from baseline to 2-weeks follow-up after intervention
  Children's performance on the Unstructured Imitation Assessments (score 0-20)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Lense, Principal Investigator — Vanderbilt University Medical Center; Warren Jones, Principal Investigator — Emory University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States